CLINICAL TRIAL: NCT04800536
Title: Cardiovascular Effects of Rapidly Declining Plasma Glucose in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-20033627
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
Keywords: Plasma glucose decline rate; Cardiovascular disease; Sudden cardiac death; Glycaemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiovascular effects of rapidly declining plasma glucose (Experimental): A combined hyperglycaemic and euglycaemic clamp with a rapidly declining plasma glucose (>0.15 mmol/l/min). Plasma glucose will be measured every 5 minute and cardiovascular effects of the plasma glucose decline rate will be assessed using Holter-ECG, echocardiography, thrombelastography and blood sampling.
  Interventions: Other: Rapidly declining plasma glucose
- Cardiovascular effects of slowly declining plasma glucose (Experimental): A combined hyperglycaemic and euglycaemic clamp with slowly declining plasma glucose (<0.085 mmol/l/min). A combined hyperglycaemic and euglycaemic clamp with a slowly declining plasma glucose (>0.15 mmol/l/min). Plasma glucose will be measured every 5 minute and cardiovascular effects of the plasma glucose decline rate will be assessed using Holter-ECG, echocardiography, thrombelastography and blood sampling.
  Interventions: Other: Slowly declining plasma glucose

INTERVENTIONS:
Other: Rapidly declining plasma glucose — Acute plasma glucose decline, divided into the following three phases: 1) Hyperglycaemic phase (plasma glucose 15 mmol/l), 2) Rapid plasma glucose decline phase and 3) Euglycaemic phase (plasma glucose 4.5-5.5 mmol/l).
  Arms: Cardiovascular effects of rapidly declining plasma glucose
Other: Slowly declining plasma glucose — Acute plasma glucose decline, divided into the following three phases: 1) Hyperglycaemic phase (plasma glucose 15 mmol/l), 2) Slow plasma glucose decline phase and 3) Euglycaemic phase (plasma glucose 4.5-5.5 mmol/l).
  Arms: Cardiovascular effects of slowly declining plasma glucose

SUMMARY:
Type 1 diabetes (T1D) is an autoimmune metabolic disease characterised by impaired lack of endogenous insulin causing elevated plasma glucose levels and increased risk of microvascular and macrovascular complications. With respect to the cardiovascular system, patients with T1D have an up to 10-fold increased risk of sudden cardiac death compared to healthy individuals. Furthermore, diabetes constitutes a hypercoagulable state, which to some extent may explain why cardiovascular disease still is a major cause of mortality in patients with T1D. Due to treatment with exogenously delivered insulin, glycaemic variability with intra-day and inter-day plasma glucose concentrations fluctuating between high levels (peaks) and low levels (nadirs), are inevitable in patients with T1D. A potentially important factor in development of cardiovascular disease, associated with glycaemic variability, is the rate of increase and/or decline of plasma glucose. The aim of this study is to test the hypothesis that a rapid plasma glucose decline from a hyperglycaemic level to an euglycaemic level can induce changes in QT-interval and blood coagulation in a proarrhythmogenic and prothrombotic way.

Twenty patients with T1D with a 1:1 distribution with chronic hyperglycaemia (HbA1C ≥63 mmol/mol) and with well-controlled diabetes (HbA1C ≤53 mmol/mol) will be recruited for a crossover study including two test days (protocols), P-rapid, a combined hyperglycaemic and euglycaemic clamp with rapidly declining plasma glucose and P-slow, a combined hyperglycaemic and euglycaemic clamp with slowly declining plasma glucose. Patients will be randomised 1:1 to start with P-rapid or P-slow. The cardiovascular effects will be investigated using Holter-ECG, Thrombelastography, Echocardiography and blood sampling.

Given that cardiovascular disease is a major cause of death in patients with T1D and that patients with diabetes may be more susceptible for cardiac arrhythmias and thrombotic events compared to healthy individuals, it is important to identify cardiovascular risk factors related to acute changes in plasma glucose in order to improve prevention strategies and therapy.

ELIGIBILITY:
Inclusion criteria - chronic hyperglycaemia cohort

* Informed and written consent
* Type 1 diabetes
* Age ≥18 years
* C-peptide negative (<0.2 nmol/l)
* Insulin treatment for ≥1 year
* HbA1C ≥63 mmol/mol

Inclusion criteria - well-controlled cohort

* Informed and written consent
* Type 1 diabetes
* Age ≥18 years
* C-peptide negative (<0.2nmol/l)
* Insulin treatment for ≥1 year
* HbA1C ≤53 mmol/mol

Exclusion criteria - both cohorts

* Arrhythmia diagnosed prior to or at the time of the screening visit
* ECG with left or right bundle branch block diagnosed prior to the screening visit.
* Implantable cardioverter defibrillator or pacemaker at the time of inclusion
* Heart failure diagnosed prior to the screening visit (left ventricular ejection fraction < 45%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated myxoedema)
* Anaemia (male: haemoglobin <8.0 mmol/l; female: haemoglobin <7.0 mmol/l)
* Treatment with anticoagulant or antiplatelet treatment
* Bleeding disorder diagnosed prior to the screening visit

Withdrawal criteria

• The participants may withdraw at will at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
QTc interval | 0-255 minutes
  Difference in mean QTc (ms) interval from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.

SECONDARY OUTCOMES:
Cardiac function | 0-255 minutes
  Difference in ventricular systolic function (measured by echocardiography) from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.
Heart rate variability | 0-255 minutes
  Difference in the sympathetic/parasympathetic balance (measured by heart rate variability) during a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.
Haemostatic balance | 0-255 minutes
  Difference in activation of coagulation and fibrinolysis (measured by TEG) from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.
Endothelial activation and damage | 0-255 minutes
  Difference in endothelial activation and damage (measured by Syndecan-1, Soluble thrombomodulin and sVE-cadherin) (ng/ml) from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.
Plasma glucose decline rate and counterregulatory hormonal response | 0-255 minutes
  Difference in counterregulatory hormonal response (plasma glucagon, catecholamines, cortisol, and growth hormone) from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.
Plasma glucose decline rate and oxidative stress | 0-255 minutes
  Difference in vascular oxidative stress (Tetrahydrobiopterin/dihydrobiopterin ratio, Dehydroascorbic acid/Ascorbic acid ratio, Asymmetric dimethylarginine/Arginine ratio, Malondialdehyde) from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.
Plasma glucose decline rate and potassium | 0-255 minutes
  Difference in plasma potassium concentration during a rapid plasma glucose decline compared to a slow plasma glucose decline from a hyperglycaemic level to an euglycaemic level.
Plasma glucose decline rate and symptomatic response | 0-255 minutes
  Difference in symptomatic response (Edinburgh hypoglycaemia symptom scale) from a hyperglycaemic level to an euglycaemic level preceded by a rapid plasma glucose decline compared to a slow plasma glucose decline in patients with T1D with chronic hyperglycaemia and well-controlled diabetes, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen - Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No